CLINICAL TRIAL: NCT05116774
Title: A Randomized, Open-Label, Multicenter, Parallel-Group Study to Evaluate the Efficacy, Safety, and Tolerability of Oral BCX9930 Monotherapy for the Treatment of Paroxysmal Nocturnal Hemoglobinuria in Subjects With Inadequate Response to C5 Inhibitor Therapy
Brief Title: BCX9930 for the Treatment of Paroxysmal Nocturnal Hemoglobinuria (PNH) in Participants With Inadequate Response to C5 Inhibitor Therapy
Acronym: REDEEM-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCX9930-202; 2020-004438-39 (EudraCT Number)
Record Dates: First submitted 2021-11-02; First posted 2021-11-11 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
Keywords: BCX9930; factor D inhibitor; proximal complement inhibitor; oral therapy; paroxysmal nocturnal hemoglobinuria; inadequate response to C5 inhibitor; C5 inhibitor; eculizumab; ravulizumab
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — eculizumab; ravulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BCX9930/BCX9930 (Experimental): Participants were randomized to receive BCX9930 during Part 1 and continued to receive the same during Part 2. Per protocol amendment, participants who previously received 500 mg twice daily (BID) and remained on study treatment were dose adjusted to 400 mg BID. For all newly enrolled participants, at the initiation of BCX9930 dosing, participants were administered a dose of 200 mg BID for the first 14 days of treatment before increasing to 400 mg BID. The maximum treatment duration on BCX9930 in Part 1 was 24 weeks. The overall maximum treatment duration on BCX9930 was 377 days.
  Interventions: Drug: BCX9930
- C5-Inhibitor (C5-INH)/BCX9930 (Active Comparator): Participants randomized to this group continued the existing C5-INH therapy during Part 1. After the sponsor decided to halt enrolment in the study permanently and terminate the study, participants entered Part 2 where they switched to open-label BCX9930 monotherapy prior to Week 24, if earlier. The maximum treatment duration on C5-INH in Part 1 was 24 weeks. The maximum treatment duration on BCX9930 was 197 days.
  Interventions: Drug: Eculizumab; Drug: Ravulizumab; Drug: BCX9930

INTERVENTIONS:
Drug: Eculizumab — Administered by intravenous infusion per current dose regimen
  Other Names: Soliris
  Arms: C5-Inhibitor (C5-INH)/BCX9930
Drug: Ravulizumab — Administered by intravenous infusion per current dose regimen
  Other Names: Ultomiris, ALXN1210, ravulizumab-cwvz
  Arms: C5-Inhibitor (C5-INH)/BCX9930
Drug: BCX9930 — Administered orally twice daily

SUMMARY:
The purpose of this study was to determine the efficacy and safety of BCX9930 monotherapy for the treatment of PNH compared to continued C5 inhibitor therapy in adult PNH participants with residual anemia despite treatment with a C5 inhibitor.

DETAILED DESCRIPTION:
This was a randomized, active comparator-controlled, open-label, parallel-group, 2-part study. Parts 1 and 2 were conducted in the same participants.

Part 1 of the study was designed to evaluate the efficacy, safety, and tolerability of oral BCX9930 monotherapy for 24 weeks versus continuing C5 inhibitor therapy in participants with PNH with inadequate response to their current C5 inhibitor therapy. Participants were randomized to either discontinue C5 inhibitor therapy and start BCX9930 monotherapy or to continue C5 inhibitor therapy for the 24-week randomized treatment period. The primary efficacy and safety analyses were based on Part 1.

Part 2 of the study was designed to evaluate the long-term safety, tolerability, and effectiveness of BCX9930 monotherapy when administered through Week 52. All participants in Part 2 received BCX9930. Participants who were randomized to BCX9930 monotherapy in Part 1 continued to receive BCX9930 in Part 2. Participants who were randomized to C5 inhibitor therapy in Part 1 discontinued that therapy at the Week 24 visit and received BCX9930 in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥ 18 years old
* Body weight ≥ 40 kg
* Documented diagnosis of PNH
* Currently being treated with a stable C5 inhibitor regimen
* Documentation of current vaccinations against Neisseria meningitidis and Streptococcus pneumoniae or willing to start vaccination series
* At screening: PNH clone size of ≥ 10% and hemoglobin ≤ 10.5 g/dL

Exclusion Criteria:

* Known history of or existing diagnosis of hereditary complement deficiency
* History of hematopoietic cell transplant or solid organ transplant or anticipated candidate for transplantation
* Myocardial infarction or cerebrovascular accident within 30 days prior to screening, or current and uncontrolled clinically significant cardiovascular or cerebrovascular condition
* History of malignancy within 5 years prior to the screening visit
* Active bacterial, viral, or fungal infection or any other serious infection within 14 days prior to screening
* Treatment with anti-thymocyte globulin within 180 days prior to screening
* Initiation of treatment with an erythrocyte or platelet growth factor, or danazol within 28 days prior to screening
* Receiving iron supplementation with an unstable dose in the 28 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Austin G Kulasekararaj, MBBS, MD, Principal Investigator — King's College Hospital NHS Trust
Locations (7):
- Investigative Site, Paris, France
- Investigative Site, Budapest, Hungary
- Investigative Site, Rome, Italy
- Spain (2):
  - Investigative Site, Barcelona
  - Investigative Site, Valencia
- United Kingdom (2):
  - Investigative Site, Leeds
  - Investigative Site, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total 12 participants were randomized and treated.
Pre-assignment Details: The study was conducted in France, Hungary, Italy, Spain and United Kingdom.
Groups:
- BCX9930/BCX9930: Participants were randomized to receive BCX9930 during Part 1 and continued to receive the same during Part 2. Per protocol amendment, participants who previously received 500 mg twice daily (BID) orally and remained on study treatment were dose adjusted to 400 mg BID. For all newly enrolled participants, at the initiation of BCX9930 dosing, participants were administered a dose of 200 mg BID for the first 14 days of treatment before increasing to 400 mg BID. The maximum treatment duration on BCX9930 in Part 1 was 24 weeks. The overall maximum treatment duration on BCX9930 was 377 days.
Period: Part 1 (up to 24 Weeks)
Arm/Group | BCX9930/BCX9930 | C5-Inhibitor (C5-INH)/BCX9930
Started | 8 | 4
Completed | 7 | 3
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 1 | 0
Period: Part 2 (up to 52 Weeks)
Arm/Group | BCX9930/BCX9930 | C5-Inhibitor (C5-INH)/BCX9930
Started | 7 | 3
Completed | 3 | 2
Not Completed | 4 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Miscellaneous | 3 | 1

BASELINE CHARACTERISTICS:
Population: The safety population included all participants who received at least 1 dose of study drug, whether C5 inhibitor or BCX9930.
Groups:
- BCX9930/BCX9930: Participants were randomized to receive BCX9930 during Part 1 and continued to receive the same during Part 2. Per protocol amendment, participants who previously received 500 mg BID and remained on study treatment were dose adjusted to 400 mg BID. For all newly enrolled participants, at the initiation of BCX9930 dosing, participants were administered a dose of 200 mg BID for the first 14 days of treatment before increasing to 400 mg BID. The maximum treatment duration on BCX9930 in Part 1 was 24 weeks. The overall maximum treatment duration on BCX9930 was 377 days.
- C5-INH/BCX9930: Participants randomized to this group continued the existing C5-INH therapy during Part 1. After the sponsor decided to halt enrolment in the study permanently and terminate the study, participants entered Part 2 where they switched to open-label BCX9930 monotherapy prior to Week 24, if earlier. The maximum treatment duration on C5-INH in Part 1 was 24 weeks. The maximum treatment duration on BCX9930 was 197 days.
- Total: Total of all reporting groups
Arm/Group | BCX9930/BCX9930 | C5-INH/BCX9930 | Total
Number analyzed (Participants) | 8 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (17.66) | 48.5 (14.25) | 55.3 (16.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 4 | 1 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 2 | 7
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 5 | 2 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Change From Baseline in Hemoglobin at Week 24
Time Frame: Baseline, Week 24
Population: Participants in the all subjects as treated (ASaT) population in Part 1 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Groups:
- BCX9930: Participants were randomized to receive BCX9930 during Part 1. Per protocol amendment, participants who previously received 500 mg BID and remained on study treatment were dose adjusted to 400 mg BID. For all newly enrolled participants, at the initiation of BCX9930 dosing, participants were administered a dose of 200 mg BID for the first 14 days of treatment before increasing to 400 mg BID. The maximum treatment duration on BCX9930 in Part 1 was 24 weeks.
- C5-INH: Participants randomized to this group continued the existing C5-INH therapy during Part 1. The maximum treatment duration on C5-INH in Part 1 was 24 weeks.
Arm/Group | BCX9930 | C5-INH
Number analyzed (Participants) | 8 | 4
grams per deciliter (g/dL)
  Baseline | 9.12 (1.096) | 9.13 (0.847)
  Change at Week 24: number analyzed (Participants) | 6 | 2
  Change at Week 24 | 3.48 (0.674) | 0.72 (0.884)

2. Secondary Outcome: Part 1: Number of Participants Who Were Transfusion-free
Description: The number of participants who did not receive any transfusions (packed red blood cells [pRBCs] or whole blood) during the period of interest were reported. Participants who were transfusion free were defined for each treatment group as the number of participants who did not receive any transfusions (pRBCs or whole blood) during the period of interest from the start to the end, inclusive, divided by the total number of participants in that treatment group at the start of the period of interest. Participants who (1) discontinued treatment prior to Week 24, or (2) did not receive a transfusion during the period of interest despite recording a hemoglobin (Hb) value ≤ 9 g/dL with symptoms assessed by the investigator as warranting transfusion or a Hb value ≤ 7 g/dL regardless of symptoms were not considered transfusion free.
Time Frame: From Week 4 to Week 24
Population: Participants in the ASaT population in Part 1 were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | BCX9930 | C5-INH
Number analyzed (Participants) | 8 | 4
Participants | 7 | 4

3. Secondary Outcome: Part 1: Number of Units of pRBCs Transfused
Time Frame: From Week 4 to Week 24
Population: Participants in the ASaT population in Part 1 were analyzed.
Measure: Number; unit: units of pRBCs
Arm/Group | BCX9930 | C5-INH
Number analyzed (Participants) | 8 | 4
units of pRBCs | 0 | 0

4. Secondary Outcome: Part 1: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Scale Score
Description: The FACIT-Fatigue scale questionnaire was used to determine the level of fatigue experienced by participants. This questionnaire was a 13-item measure that assessed self-reported fatigue and its impact upon daily activities and function. Item scores ranged from 0 ("not at all") to 4 ("very much"), and the total score ranged from 0 to 52, with higher scores indicating greater quality of life.
Time Frame: Baseline, Week 24
Population: Participants in the ASaT population in Part 1 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | BCX9930 | C5-INH
Number analyzed (Participants) | 6 | 2
Scores on a scale
  Baseline | 36.3 (9.69) | 40.0 (8.49)
  Change at Week 24: number analyzed (Participants) | 3 | 1
  Change at Week 24 | -0.3 (12.86) | 1.0

5. Secondary Outcome: Part 1: Percent Change From Baseline in Lactate Dehydrogenase
Time Frame: Baseline, Week 24
Population: Participants in the ASaT population in Part 1 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- C5-INH: Participants randomized to this group continued the existing C5 INH therapy during Part 1. The maximum treatment duration on C5-INH in Part 1 was 24 weeks.
Arm/Group | BCX9930 | C5-INH
Number analyzed (Participants) | 7 | 2
percent change | 24.3 (53.07) | -21.0 (4.03)

6. Secondary Outcome: Part 1: Percentage (%) Reduction in the Rate of pRBC Units Transfused
Description: The rate of pRBC units transfused from Week 4 to Week 24 was calculated and compared to the rate of pRBC units transfused prestudy during the 12 months prior to screening. The percent reduction in rate of pRBC units transfused was the percent difference in rate relative to the prestudy rate, calculated as: (current rate - prestudy rate)/prestudy rate * 100%. Total rate among all participants was evaluated here. Rate of pRBC units transfusion was defined as the percentage of participants who received pRBC transfusions.
Time Frame: Prestudy (12 months prior to screening) and from Week 4 to Week 24
Population: Participants in the ASaT population in Part 1 were analyzed.
Measure: Number; unit: percent reduction
Arm/Group | BCX9930 | C5-INH
Number analyzed (Participants) | 8 | 4
percent reduction | 100 | NA — No participants received pRBC transfusion at pre-study in the "C5-INH" arm, and therefore the percentage reduction, based on the formula provided, was not calculable.

7. Secondary Outcome: Part 1: Number of Participants With Hemoglobin ≥ 12 Grams Per Deciliter (g/dL)
Time Frame: Week 24
Population: Participants in the ASaT population in Part 1 with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | BCX9930 | C5-INH
Number analyzed (Participants) | 6 | 4
Participants | 6 | 0

8. Secondary Outcome: Part 1: Number of Participants Who Achieved Hemoglobin Stabilization
Description: Hemoglobin stabilization was defined as the participants who avoided 2 g/dL or greater decrease in hemoglobin in the absence of transfusion from Week 4 to Week 24.
Time Frame: From Week 4 to Week 24
Population: Participants in the ASaT population in Part 1 with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | BCX9930 | C5-INH
Number analyzed (Participants) | 5 | 4
Participants | 5 | 4

9. Secondary Outcome: Part 1: Change From Baseline in Complement Component 3 (C3)-Opsonized Red Blood Cells (RBCs)
Description: Red blood cells opsonized by C3 were to be assessed by flow cytometry .
Time Frame: Baseline, Week 24
Population: No data was collected for this endpoint.
Arm/Group | BCX9930 | C5-INH
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Part 1: Change From Baseline in Total Paroxysmal Nocturnal Hemoglobinuria (PNH) RBC Clone Size
Description: The total PNH RBC clone size refers to the percentage of PNH affected (ie, Type 2 and 3) RBC cells within the total RBC population.
Time Frame: Baseline, Week 24
Population: Participants in the ASaT population in Part 1 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: % of PNH-RBC within total RBC population
Groups:
- BCX9930: Participants were randomized to receive BCX9930 during Part 1. Per protocol amendment, participants who previously received 500 mg BID and remained on study treatment were dose adjusted to 400 mg BID. For all newly enrolled participants, at the initiation of BCX9930 dosing, participants were administered a dose of 200 mg BID for the first 14 days of treatment before increasing to 400 mg BID. The maximum treatment duration on BCX9930 in Part 1 was 377 days.
Arm/Group | BCX9930 | C5-INH
Number analyzed (Participants) | 6 | 3
% of PNH-RBC within total RBC population
  Baseline | 80.51 (16.94) | 83.40 (14.34)
  Change at Week 24: number analyzed (Participants) | 3 | 2
  Change at Week 24 | 23.18 (11.81) | -6.34 (8.986)

11. Secondary Outcome: Part 1: Change From Baseline in Ratio of Total PNH RBC Clone Size to PNH White Blood Cell (WBC) Clone Size
Description: The total PNH RBC clone size refers to the percentage of PNH affected (ie, Type 2 and 3) RBCs within the total RBC population. The PNH WBC clone size refers to the percentage of PNH-affected WBCs within the total WBC population. The ratio of total PNH RBC clone size to PNH WBC clone size = ratio of percent total PNH RBCs / percent PNH WBCs.
Time Frame: Baseline, Week 24
Population: Participants in the ASaT population in Part 1 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | BCX9930 | C5-INH
Number analyzed (Participants) | 4 | 2
ratio
  Baseline | 0.8128 (0.16528) | 0.9059 (0.12113)
  Change at Week 24: number analyzed (Participants) | 3 | 2
  Change at Week 24 | 0.2336 (0.11595) | -0.0668 (0.09462)

12. Secondary Outcome: Part 1: Change From Baseline in Absolute Reticulocyte Count (ARC)
Time Frame: Baseline, Week 24
Population: Participants in the ASaT population in Part 1 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: 10^6 cells/microliter (μL)
Arm/Group | BCX9930 | C5-INH
Number analyzed (Participants) | 7 | 4
10^6 cells/microliter (μL)
  Baseline | 0.2933 (0.10453) | 0.3129 (0.16201)
  Change at Week 24: number analyzed (Participants) | 6 | 4
  Change at Week 24 | -0.2142 (0.05384) | -0.0462 (0.01823)

13. Secondary Outcome: Part 1: Number of Participants With ARC in the Normal Range
Description: Number of participants with ARC in the normal range (0.03 - 0.12 10^6 cells/uL) were reported.
Time Frame: Week 24
Population: Participants in the ASaT population in Part 1 with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | BCX9930 | C5-INH
Number analyzed (Participants) | 6 | 4
Participants | 4 | 1

14. Secondary Outcome: Part 1: Change From Baseline in Haptoglobin
Time Frame: Baseline, Week 24
Population: Participants in the ASaT population in Part 1 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | BCX9930 | C5-INH
Number analyzed (Participants) | 7 | 4
grams per liter (g/L)
  Baseline | 0.126 (0.0732) | 0.105 (0.0268)
  Change at Week 24 | -0.024 (0.0409) | -0.015 (0.0268)

15. Secondary Outcome: Part 1: Number of Participants With Haptoglobin ≥ Lower Limit of Normal (LLN) Reference Range
Description: Number of Participants With Haptoglobin ≥ LLN Reference Range (≥0.3 g/L) were reported.
Time Frame: Week 24
Population: Participants in the ASaT population in Part 1 with available data were analyzed.
Measure: Count of Participants; unit: Participants
Groups:
- BCX9930: Participants were randomized to receive BCX9930 during Part 1. Per protocol amendment, participants who previously received 500 mg BID and remained on study treatment were dose adjusted to 400 mg BID. For all newly enrolled participants, at the initiation of BCX9930 dosing, participants were administered a dose of 200 mg BID for the first 14 days of treatment before increasing to 400 mg BID. The maximum treatment duration on BCX9930 in Part 1was 24 weeks.
Arm/Group | BCX9930 | C5-INH
Number analyzed (Participants) | 7 | 4
Participants | 0 | 0

16. Secondary Outcome: Part 1: Change From Baseline in Total Bilirubin
Time Frame: Baseline, Week 24
Population: Participants in the ASaT population in Part 1 with available data were analyzed.
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | BCX9930 | C5-INH
Number analyzed (Participants) | 7 | 4
milligram per deciliter (mg/dL)
  Baseline | 3.44 (3.679) | 1.10 (0.424)
  Change at Week 24 | -2.66 (3.672) | -0.02 (0.250)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 407
Description: The safety population included all participants who received at least 1 dose of study drug, whether C5 inhibitor or BCX9930.
Groups:
- C5-INH: Participants randomized to this group continued the existing C5-INH therapy during Part 1. The maximum treatment duration on C5-INH was 24 weeks.
- BCX9930 After C5-INH: Participants who were initially randomized to continue C5-INH therapy received BCX9930 monotherapy after they had completed 24 weeks on C5-INH, or earlier after the date when sponsor decided to halt enrolment in the study permanently and terminate the study. Initially participants were to receive BCX9930 500 mg BID orally. Per protocol amendment, participants who previously received 500 mg BID and remained on study treatment were dose adjusted to 400 mg BID. For all newly enrolled participants, at the initiation of BCX9930 dosing, participants were administered a dose of 200 mg BID for the first 14 days of treatment before increasing to 400 mg BID. The maximum treatment duration on BCX9930 was 197 days.
Arm/Group | BCX9930/BCX9930 | C5-INH | BCX9930 After C5-INH
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 2/8 | 0/4 | 1/3
Other Adverse Events (participants affected / at risk) | 7/8 | 3/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCX9930/BCX9930 (N=8) | C5-INH (N=4) | BCX9930 After C5-INH (N=3)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BCX9930/BCX9930 (N=8) | C5-INH (N=4) | BCX9930 After C5-INH (N=3)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (4) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 3 (4) | 0 (0)
Fatigue (General disorders) | 3 (5) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (6) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Axillary mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (3) | 0 (0) | 0 (0)
Haemoglobinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic cytolysis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Prothrombin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The sponsor decided to terminate the development program (including this study).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT05116774/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/74/NCT05116774/SAP_001.pdf